CLINICAL TRIAL: NCT02562404
Title: Vagus Nerve Injury Post Radiofrequency Catheter Ablation for Atrial Fibrillation (Vagus Nerve Study)
Brief Title: Vagus Nerve Injury Post Radiofrequency Catheter Ablation for Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 1025037
Record Dates: First submitted 2015-09-25; First posted 2015-09-29 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2016-06

CONDITIONS: Atrial Fibrillation; Gastrointestinal Tract; Radiofrequency Catheter Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is an observational study designed to determine the extent of gastrointestinal (GI) post-procedure complications after Radiofrequency Catheter Ablation (RFCA) for atrial fibrillation (AF). This exploratory study will evaluate patient symptoms prior to the RFCA procedure, at 1 month post RFCA procedure, and at 3 months post RFCA procedure, through the administration of a questionnaire. The purpose of this study is to determine if vagus nerve injury resulting from RFCA for AF increases the risk of post-procedure GI complications that may present as temporary or permanent symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a verified medical history of atrial fibrillation.
* Male or female >18 years of age.
* Patients scheduled for an RFCA procedure, subsequent to failure of one Antiarrhythmic Drug (AAD class I, III or IV), or ablation.
* Ability to answer questions posed by the questionnaire.
* Ability to understand and sign a written informed consent form, which must be obtained prior to initiation of any study procedures.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Atrial fibrillation patients at the Intermountain Medical Center Heart Rhythm Clinic who are candidates for Radiofrequency Catheter Ablation (RFCA) will be screened for participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Symptoms Associated with Vagus Nerve Injury | At RFCA procedure, 1 month post RFCA procedure, 3 months post RFCA procedure
  The composite of symptoms associated with vagus nerve injury: increased heart rate, bloating, early satiety, heartburn, changes in bowel habits, weight loss, problems with swallowing, nausea and vomiting. These symptoms will be discovered through the administration of a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: T. Jared Bunch, MD, Principal Investigator — Intermountain Medical Center
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States